CLINICAL TRIAL: NCT05458024
Title: Randomized Controlled Trial of Vitamin D to Reduce Racial Disparity in Chronic Pain Following Motor Vehicle Collision
Brief Title: Vitamin D to ENhance TraUma REcovery
Acronym: VENTURE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21-2589; R21MD016467 (NIH)
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2023-05

CONDITIONS: Musculoskeletal Pain
Keywords: Vitamin D; Motor Vehicles; Pain; Racial Disparity
MeSH Terms: conditions — Musculoskeletal Pain; Pain | interventions — Ergocalciferols

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial enrolling motor vehicle collision survivors within 24 hours after injury (n=90, 45 non-Hispanic Black, and 45 non-Hispanic White) will be randomized in 1:1 allocation of a one-time dose of either Vitamin D or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a blinded study. Investigators, participants, and coordinators will be blinded to the treatment assignment. Active and placebo treatments will be indistinguishable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ergocalciferol (Vitamin D2) (Active Comparator): 300,000 international units (IUs) of Ergocalciferol in 6 50,000 IU capsules. These will be given in a single dose prior to discharge from the Emergency Department.
  Interventions: Drug: Vitamin D 2
- Ergocalciferol placebo (Placebo Comparator): Inert substance will be administered in 6 capsules indistinguishable from the 50,000 IU Ergocalciferol capsules administered in the active treatment arm.
  Interventions: Drug: Vitamin D2 Placebo

INTERVENTIONS:
Drug: Vitamin D 2 — 300,000 international units (IUs) of Ergocalciferol in 6 50,000 IU capsules.
  Other Names: Ergocalciferol 300,000 IU
  Arms: Ergocalciferol (Vitamin D2)
Drug: Vitamin D2 Placebo — Inert substance will be administered in 6 capsules indistinguishable from the 50,000 IU
  Other Names: Ergocalciferol Placebo
  Arms: Ergocalciferol placebo

SUMMARY:
The main objective of this study is to determine whether the administration of a single dose of Vitamin D in the Emergency Department following a motor vehicle collision can improve musculoskeletal pain severity as well as reduce musculoskeletal pain outcome disparity between Blacks and White following a motor vehicle collision. This randomized controlled trial is a pilot study to determine feasibility and potential efficacy (response to study drug, ability to reduce racial disparity in pain outcomes). This data can be used to adequately power a larger randomized controlled trial to fully assess efficacy.

DETAILED DESCRIPTION:
Motor vehicle collisions (MVCs) are one of the most common traumatic stress exposures in the US, and the most common for which individuals seek emergency department (ED) care. More than 1 million Black Americans (Blacks) come to the ED after MVC each year, and >90% of such ED MVC patients are discharged home with a diagnosis of acute musculoskeletal pain (MSP)/strain only. More than 80% of these individuals report acute moderate or severe (mod/sev) MSP in the ED, and >50% of those with acute mod/sev MSP transition to chronic MSP. MVCs, as well as pain after MVC, disproportionately affect Blacks vs. Whites. For example, in previous cohort studies 67% of Blacks had mod/sev MSP six months after MVC, vs. only 40% of Whites. Interventions are urgently needed that prevent chronic MSP and reduce these MSP outcome disparities.

One safe, inexpensive, widely available, and well-tolerated intervention, with exciting potential to achieve these goals, is Vitamin D (Vitamin D). The dose of Ergocalciferol that the investigators propose, 300,000 IU, has been shown to effectively raise Vitamin D concentration by ~9 ng/ml, and to raise serum 25 hydroxyvitamin D concentration above 30 ng/ml (Vitamin D sufficient levels) for over 3 months5. The ability of this single-dose protocol to raise Vitamin D will be a primary feasibility endpoint of this pilot study.

Importantly, this dose is extremely well-tolerated: in previous trials, reports of side effects/adverse events is rare,6 many studies administering single, high-dose regimens report no side effects7-9, and the most common side effects have been mild GI complaints (e.g. nausea).6 Vitamin D administration has also been demonstrated to be safe, even among individuals who are already Vitamin D sufficient. 10-12

Chronic pain is associated with reduced mental and physical health and interferes with essential activities of daily life. Currently there are limited treatment options to address chronic pain once it has become established and the overarching aim of this clinical trial is to prevent chronic pain development, therefore there is a critical unmet need of safe, non-addictive, non-invasive preventative treatment options that can be administered to MVC survivors in the aftermath of an injury. This study has the potential to benefit participants and future MVC survivors and improve pain and general health outcomes. The risks of taking Vitamin D are small. Side effects from Vitamin D are rare, however, it is possible that over supplementation of Vitamin D may be associated with headache, loss of appetite, dry mouth, metallic taste, and nausea/vomiting.

Primary Objective:

1. Assess the feasibility of the Randomized Controlled Trial (RCT) protocol by (a) calculating recruitment rate and participant retention, and (b) measuring the ability of Vitamin D administration to generate sustained increases in whole-blood Vitamin D concentrations (assessed 3 months after MVC).
2. To demonstrate the preliminary efficacy of Vitamin D administration per protocol on decreasing overall MSP severity during the 3 months following MVC, and reducing MSP outcome disparity between Blacks and Whites following MVC.

Secondary Objectives:

The investigators will assess the effect of race and sex on treatment outcomes in secondary analyses. This will be accomplished using two analytic strategies. First, a sex X treatment interaction term (secondary analyses) will be entered into the statistical models to assess pain reduction in response to treatment. Second, a stratified analysis will be performed which will examine the influence of both sex and race on treatment effect on primary and secondary outcomes. Further, Secondary stratified analyses evaluate the influence of initial vitamin D level on treatment response. In addition, exploratory analyses on the relationship of vitamin D outcome and trajectory of pain as well as restricting analyses to participants with vitamin D deficiency at baseline will be performed. Secondary analyses will examine treatment effects adjusting for any baseline differences in psychosocial factors between treatment arms.

Long-Term Aims Beyond the Present Proposal:

To use data collected to design and adequately power a larger-scale RCT assessing the efficacy of Vitamin D treatment in decreasing chronic pain in high-risk patients presenting for treatment in the aftermath of MVC and to reduce racial disparity in pain outcomes following MVC.

Described the sequence of events in recruiting 90 patients in a multi-center randomized controlled trial. To assess a key primary outcome, 50% white and 50% black MVC will be enrolled into the study. Each participant will be screened in based on a point of care Vitamin D test. This will be performed at the time of screening. Individuals with a Vitamin D level <100 ng/ml will be enrolled. Patients will be randomized 1:1 to receive a single dose of 300,000 IU of ergocalciferol versus placebo and followed for 3 months. At 3 months, patients will send a blood sample easily collected at home on a blood spot card to assess Vitamin D level 3 months following injury which is a key feasibility primary outcome.

Patients presenting to the ED within 24 hours of MVC (n=90, 45 non-Hispanic Black, and 45 non-Hispanic White) will receive a single dose of study drug prior to ED discharge (1:1 allocation 300,000 IU ergocalciferol or placebo). Prior to study drug administration, a baseline assessment will be performed (see below), and a fingerstick blood sample will be obtained to evaluate 25-hydroxyvitamin D level. Telephone follow-ups assessing primary and secondary outcomes and potential adverse events will be performed 3 weeks, 6 weeks, and 3 months after ED enrollment by study Research Assistants using web-based REDCap™ software. At 3 months, participants will also perform fingerstick blood collection at home and mail to the study team to enable assessment of 3 month 25-hydroxyvitamin D concentration by treatment group.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years and ≤ 65 years of age
* Admitted to ED within 24 hours of motor vehicle collision
* Plan to discharge to home from the emergency department
* Stated willingness to comply with all study procedures and availability for the duration of the study (with the exception of the blood draw sample collected in the ED, which is optional)
* Has a smartphone with continuous service >1 year
* Able to speak and read English
* Alert and oriented, and capable of engaging in informed consent
* Willing to take on-time dose of study medication (6 capsules of Vitamin D or placebo)
* Non-Hispanic white or non-Hispanic black
* Point of care Vitamin D level <100 ng/ml
* During ED admission pain severity must be at least 4/10 or higher

Exclusion Criteria:

* Substantial comorbid injury (e.g., long bone fracture)
* Pregnancy/breastfeeding
* Prisoner status
* Chronic daily opioid use prior to MVC (>20 mg oral daily morphine equivalents)
* Active psychosis, suicidal ideation, or homicidal ideation
* Plans for hospital admission
* Known chronic kidney disease, stage 4 or higher (GFR≤29)
* Intubated and sedated at time of enrollment
* Inability to provide informed consent (receipt of sedative, hypnotic agent making the patient non-decisional for consent)
* Vitamin D supplements in excess of 800 IU daily
* Any other history or condition that would, in the site investigator's judgement, indicate that the patient would very likely be non-compliant with the study or unsuitable for the study (e.g., might interfere with the study, confound interpretation, or endanger patient)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel McLean, Principal Investigator — University of North Carolina, Chapel Hill
Locations (4):
- United States (4):
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared on request provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina (UNC).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 12 months following publication and continuing for 36 months
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants presented to participating emergency departments after a motor vehicle collision. The first participant was enrolled on January 24, 2023 and the last participant was enrolled January 30, 2024
Pre-assignment Details: Of 233 participants who were screened for eligibility, 71 were enrolled and randomized to treatment
Groups:
- Ergocalciferol (Vitamin D2): 300,000 international units (IUs) of Ergocalciferol in 6 50,000 IU capsules. These were given in a single dose prior to discharge from the Emergency Department.
- Ergocalciferol Placebo: Inert substance was administered in 6 capsules indistinguishable from the 50,000 IU Ergocalciferol capsules administered in the active treatment arm.
Period: Overall Study
Arm/Group | Ergocalciferol (Vitamin D2) | Ergocalciferol Placebo
Started | 36 | 35
Provided 3-Month Pain Data | 20 | 23
Complete 3-Month Follow Up Assessments | 24 | 28
Completed | 35 | 34
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ergocalciferol (Vitamin D2) | Ergocalciferol Placebo | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.8 (13.6) | 35.2 (13.3) | 36 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 17 | 18 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 36 | 35 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 21 | 41
  White | 16 | 14 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 35 | 71
Pain [Mean (Standard Deviation); unit: Score on a scale] — Participants rated current pain on an 11-point scale where 0 = no pain or tenderness and 10 = severe pain or tenderness. Higher scores indicate more severe pain.
  Score on a scale | 6.89 (1.97) | 6.77 (1.83) | 6.83 (1.89)
Vitamin D [Mean (Standard Deviation); unit: ng/ml] — Vitamin D levels were collected with a blood spot card in the Emergency Department.
  ng/ml | 18.2 (11.4) | 16.3 (8.85) | 17.3 (10.2)

OUTCOME MEASURES:

1. Primary Outcome: Chronic Pain Severity
Description: Estimates of efficacy will be obtained via repeated measures analysis of pain severity over the 3 months following injury using mixed effects models. Pain will be assessed using a 0-10 numeric rating scale with 0 indicating no pain and 10 indicating pain as severe as one can imagine. Higher scores represent worse outcome. These values (collected in identical fashion over 3 months following motor vehicle collision) will be entered into a linear mixed model, and overall effect estimates (beta coefficients) among treatment groups will be determined
Time Frame: Over 3 months following MVC
Population: Data are reported for all participants who had 3-month pain data available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ergocalciferol (Vitamin D2) | Ergocalciferol Placebo
Number analyzed (Participants) | 20 | 23
score on a scale
  3 week pain | 4.33 (2.81) | 5 (2.29)
  4 week pain | 4.39 (2.92) | 4.22 (2.04)
  5 week pain | 3.81 (2.80) | 3.92 (1.95)
  6 week pain | 3.29 (2.98) | 3.81 (2.48)
  3 month pain | 2.7 (2.98) | 3.0 (2.11)
Statistical Analysis 1: Comparison: Ergocalciferol (Vitamin D2) vs Ergocalciferol Placebo; Test type: Superiority; p = 0.83, Mixed Models Analysis; Beta coefficient = -.14

2. Primary Outcome: Chronic Pain Race X Treatment Arm Interaction
Description: Estimates of interaction between race and treatment assignment will be obtained via repeated measures analysis of pain severity over the 3 months following injury using mixed effects models. Pain will be assessed using a 0-10 numeric rating scale with 0 indicating no pain and 10 indicating pain as severe as one can imagine. Higher scores represent worse outcome. These values (collected in identical fashion over 3 months following burn injury) will be entered into a linear mixed model, and the beta coefficient for the race by treatment interaction term will be assessed.
Time Frame: Over 3 months following MVC
Population: Data are reported for all participants who had 3-month pain data available.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Ergocalciferol (Vitamin D2): White Participants: Non-Hispanic White participants given 300,000 international units (IUs) of Ergocalciferol in 6 50,000 IU capsules. These were given in a single dose prior to discharge from the Emergency Department.
- Ergocalciferol (Vitamin D2): Black Participants: Non-Hispanic Black participants given 300,000 international units (IUs) of Ergocalciferol in 6 50,000 IU capsules. These were given in a single dose prior to discharge from the Emergency Department.
- Ergocalciferol Placebo: White Participants: Non-Hispanic White participants given Inert substance administered in 6 capsules indistinguishable from the 50,000 IU Ergocalciferol capsules administered in the active treatment arm.
- Ergocalciferol Placebo: Black Participants: Non-Hispanic Black participants given Inert substance administered in 6 capsules indistinguishable from the 50,000 IU Ergocalciferol capsules administered in the active treatment arm.
Arm/Group | Ergocalciferol (Vitamin D2): White Participants | Ergocalciferol (Vitamin D2): Black Participants | Ergocalciferol Placebo: White Participants | Ergocalciferol Placebo: Black Participants
Number analyzed (Participants) | 10 | 10 | 9 | 14
score on a scale
  3 week pain | 3 (2) | 5.91 (2.88) | 4.3 (2.16) | 5.47 (2.33)
  4 week pain | 2.69 (2.18) | 6.60 (2.22) | 3.78 (1.86) | 4.50 (2.18)
  5 week pain | 2.23 (2.13) | 5.38 (2.53) | 2.78 (2.28) | 4.60 (1.4)
  6 week pain | 1.79 (2.04) | 4.79 (3.07) | 3.30 (2.75) | 4.13 (2.33)
  3 month pain | 1.00 (1.89) | 4.40 (2.95) | 2.56 (2.01) | 3.29 (2.20)
Statistical Analysis 1: Comparison: Ergocalciferol (Vitamin D2): White Participants vs Ergocalciferol (Vitamin D2): Black Participants vs Ergocalciferol Placebo: White Participants vs Ergocalciferol Placebo: Black Participants; Test type: Superiority; p = 0.21, Mixed Models Analysis — Analyses were adjusted for sex, baseline pain, and baseline vitamin D levels; Beta coefficient = -1.41

3. Primary Outcome: Enrollment of the 90-participant Sample Size During Enrollment Period (Feasibility)
Description: One feasibility measure of this study is demonstrating the ability to recruit 90 patients into the trial within 15 months of enrollment of the first participant. Feasibility of enrollment is defined as the number of potential participants screened for study eligibility versus the number of persons who enrolled in the study.
Time Frame: 13 months of enrollment after the first participant
Population: Although the study originally planned to enroll for a total of 15 months, due to administrative funding delays the start date was delayed resulting in a 13-month enrollment window.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants Screened: Participants who present to the participating Emergency Department after experiencing a motor vehicle collision.
Arm/Group | All Participants Screened
Number analyzed (Participants) | 233
Participants | 71

4. Primary Outcome: Percent of Participants Who Are Compliant With Follow-up (Feasibility)
Description: The primary objective of this study is to ensure that the investigators are able to make follow-up assessments on a majority of participants. The percent of participants who are compliant with follow-up will be determined 3 months following their motor vehicle collision. Feasibility is defined as >80% of enrolled participants at 3 months following Motor Vehicle Collision (MVC).
Time Frame: through study completion, 3 months following MVC
Population: Data are reported for participants who completed various follow up assessments at the end of 3 months.
Measure: Number; unit: percent of participants
Arm/Group | Ergocalciferol (Vitamin D2) | Ergocalciferol Placebo
Number analyzed (Participants) | 36 | 35
percent of participants | 66.7 | 80.0

ADVERSE EVENTS:
Time Frame: 30 days after receiving the study drug; participants received study drug within 24 hours of motor vehicle collision
Description: In addition to the clinicaltrials.gov definition, a preexisting condition was recorded as an adverse event if the frequency, intensity, or the character of the condition worsened during the study period. All unresolved adverse events were followed by the investigator until the events were resolved, the subject was lost to follow-up, or the adverse event was otherwise explained.
Arm/Group | Ergocalciferol (Vitamin D2) | Ergocalciferol Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/35
Other Adverse Events (participants affected / at risk) | 9/36 | 6/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ergocalciferol (Vitamin D2) (N=36) | Ergocalciferol Placebo (N=35)
Distressing thoughts related to MVC (Psychiatric disorders) | 6 (6) | 3 (3)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Distressing thoughts related to MVC and depression (Psychiatric disorders) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
High rate of missing Vitamin D levels at 3-months could impact findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT05458024/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-29): https://cdn.clinicaltrials.gov/large-docs/24/NCT05458024/ICF_002.pdf